CLINICAL TRIAL: NCT04333641
Title: Development of Novel Imaging Markers Predicting the Progression of Abdominal Aortic Aneurysm Using 3D Computed Tomography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0443
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: abdominal Aortic Aneurysm; CT; risk factor
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- small AAA patients: all patients with small AAA

SUMMARY:
Study purpose: This study will investigate anatomical factors associated with increased risk of major adverse aorta-related event and accelerated growth of abdominal aneurysm based on 3-dimensional analysis of CT images.

Study design: a multicenter single-arm prospective observational study.

Subject: patients with small abdominal aortic aneurysm with maximal diameter of 30-50 mm (n=323)

Methods: Patients diagnosed with small AAA based on CT will be enrolled after considering inclusion and exclusion criteria and prospectively followed clinically and with CT at 1 year.

Primary endpoint: Major adverse aorta-related events (death, aortic rupture, or aneurysm growth >0.4 cm per year) at 1 year

Secondary endpoints: 1) clinical events : death, aortic rupture, aneurysm growth >0.4 cm per year, surgical or endovascular repair 2) Changes in CT parameters of aneurysm: diameter, volume, wall shear stress

DETAILED DESCRIPTION:
Prospective single-arm multicenter registry

ELIGIBILITY:
Inclusion Criteria:

- abdominal aortic aneurysm with maximum diameter of 30-50 mm

Exclusion Criteria:

* Age <19 years
* Serum Cr> 1.5mg/dL or eGFR<30 mL/min
* Known allergic reactions to iodine contrast media
* Women in pregnancy or women of childbearing age
* Abdominal aortic aneurysms indicated for endovascular or surgical repair (symptomatic aneurysm or aneurysms with diameter >5cm)
* Saccular type aneurysm, infected or inflammatory aneurysm
* Combined aortic dissection
* Aneurysms associated with genetic or connective tissue diseases (Marfan syndrome, Shprintzen-Goldberg syndrome, Loeys-Dietz syndrome, Takayasu's arteritis, Behcet's disease)
* Past history of surgical or endovascular repair of aorta
* Any surgical or endovascular repair planned within 1 year
* Life expectancy < 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with small abdominal aortic aneurysm with maximal aneurysm of 30 ~50 mm
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Major adverse aorta-related events | 1 year
  Composite event of death, aortic rupture, or aneurysm growth >0.4 cm per year

SECONDARY OUTCOMES:
Number of clinical events | 1 year
  death, aortic rupture, aneurysm growth >0.4 cm per year, surgical or endovascular repair
Change in CT parameter of aneurysm | 1 year
  diameter
Change in CT parameter of aneurysm | 1 year
  volume
Change in CT parameter of aneurysm | 1 year
  wall shear stress

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No